CLINICAL TRIAL: NCT05741814
Title: Propofol Sedation vs. Anaesthetist Guided Anaesthesia in Oocyte Pickup - a Prospective Study
Brief Title: Propofol Sedation vs. Anaesthetist Guided Anaesthesia in Oocyte Pickup
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wunschbaby Institut Feichtinger (Other)
Responsible Party: Principal Investigator, Michael Feichtinger, Principal Investigator, Wunschbaby Institut Feichtinger
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 518-2022
Record Dates: First submitted 2022-11-07; First posted 2023-02-23 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: IVF
Keywords: Oocyte Retrieval; Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Patients receive gynaecologist guided individualised propofol sedation
  Interventions: Drug: Propofol
- Anaesthetic guided anaesthesia (Active Comparator): Patients receive anaesthetist guided full anaesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Gynecologist guided individualised propofol only sedation

SUMMARY:
Patients undergoing their first course of in vitro fertilisation receive either gynaecologist guided propofol only sedation or anaesthetist guided full anaesthesia. Patient satisfaction and clinical outcome will be evaluated afterwards.

ELIGIBILITY:
Inclusion Criteria:

Patient undergoing first oocyte pickup Understands german language to fill out questionnaire

Exclusion Criteria:

BMI >30 BMI <17 Heavy endometriosis Patients undergoing a consecutive IVF attempt

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women between 18-40 years
Enrollment: 100 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | May 2022-March 2023
  Patient satisfaction measured by the ZUF-8 questionnaire (Questionnaire to evaluate patient satisfaction)

SECONDARY OUTCOMES:
Retrieved oocytes | 1st of May 2022- 1st of March 2023
  Number of retrieved oocytes
Mature oocytes | 1st of May 2022-1st of March 2023
  Number of mature oocytes
Fertilised oocytes | 1st of May 2022- 1st of March 2023
  Number of fertilised oocytes
Cryopreserved blastocysts | 1st of May 2022- 1st of March 2023
  Number of cryopreserved blastocysts
Pregnancy rate | 1st of May 2022- 1st of March 2023
  Pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Wunschbaby Institut Feichtinger, Vienna, Austria